CLINICAL TRIAL: NCT01803841
Title: Korea Transradial Coronary Intervention Prospective Registry (KOTRI)
Acronym: KOTRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: The Korean Society of Cardiology (Other)
Responsible Party: Principal Investigator, Yoon Junghan, Professor of Cardiology, Department of Internal Medicine, Yonsei University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOTRI
Record Dates: First submitted 2013-02-25; First posted 2013-03-04 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transradial access (Active Comparator): Coronary angiography and intervention via radial artery approach
  Interventions: Procedure: Transradial coronary angiography and intervention
- Transfemoral access (Active Comparator): Coronary angiography and intervention via femoral artery approach
  Interventions: Procedure: Transfemoral coronary angiography and intervention

INTERVENTIONS:
Procedure: Transradial coronary angiography and intervention
  Arms: Transradial access
Procedure: Transfemoral coronary angiography and intervention
  Arms: Transfemoral access

SUMMARY:
The aim of this registry is to analyze several factors affecting the procedural success and clinical outcomes at 1 year of follow-up according to the approach site.

DETAILED DESCRIPTION:
This registry is a multi-center prospective registry for patients undergoing coronary angiography or percutaneous coronary intervention either transradial or transfemoral approach from 22 centers in South Korea. The aim of this registry is to analyze several factors affecting the procedural success and clinical outcomes at 1 year of follow-up according to the approach site.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive hospitalized patients undergoing coronary angiography or percutaneous coronary intervention

Exclusion Criteria:

* No exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7300 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Patient-oriented composite outcome | 1 year
  The composite of any death, non-fatal myocardial infarction, and any revascularization

SECONDARY OUTCOMES:
Access failure | Day 0 (end of procedure)
  Conversion rate of access site
Success of percutaneous coronary intervention | Day 3 (day of discharge)
  Combination of angiographic success and procedural success
  1. Angiographic success; thrombolysis in myocardial infarction (TIMI) flow grad 3 and <30% residual diameter stenosis
  2. Procedural success; Angiographic success without major procedural or in-hospital complications such as death, Q-wave myocardial infarction, or emergency bypass surgery
Procedure time | Day 0 (end of procedure)
  Procedure time according to the access site
Fluoroscopic time | Day 0 (end of procedure)
  Fluoroscopic time according to the access site

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Background] Choe JC, Cha KS, Choi JH, Kim BW, Park JS, Lee HW, Oh JH, Choi JH, Lee HC, Hong TJ, Youn YJ, Lee SH, Cho BR, Kim DI, Han KR, Jeong MH, Yoon J; Korea Transradial Coronary Intervention (KOTRI) Prospective Registry Investigators. Comparison of Frequency of Bleeding and Major Adverse Cardiac Events After Transradial Versus Transfemoral Intervention in the Recent Antiplatelet Era. Am J Cardiol. 2016 May 15;117(10):1588-1595. doi: 10.1016/j.amjcard.2016.02.033. Epub 2016 Mar 2. PMID 27026640
- [Background] Lee SH, Jeong MH, Han KR, Sim DS, Yoon J, Youn YJ, Cho BR, Cha KS, Hyon MS, Rha SW, Kim BO, Shin WY, Park KS, Cheong SS; Korean Transradial Coronary Intervention Registry Investigators. Comparison of Transradial and Transfemoral Approaches for Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome and Anemia. Am J Cardiol. 2016 May 15;117(10):1582-1587. doi: 10.1016/j.amjcard.2016.02.030. Epub 2016 Mar 2. PMID 27018932
- [Result] Youn YJ, Lee JW, Ahn SG, Lee SH, Yoon J, Cho BR, Cheong SS, Kim HY, Lee JH, Bae JH, Lee JB, Suh J, Park KS, Han KR, Jeong MH, Rha SW, Her SH, Cho YH, Kim SW. Current Practice of Transradial Coronary Angiography and Intervention: Results from the Korean Transradial Intervention Prospective Registry. Korean Circ J. 2015 Nov;45(6):457-68. doi: 10.4070/kcj.2015.45.6.457. Epub 2015 Nov 25. PMID 26617647
- See also: TRI retrospective registry electronic case report form (eCRF) — http://tricrf.medsoft.co.kr